CLINICAL TRIAL: NCT05486754
Title: Cognitive Behavioral Stress Management (CBSM) & Prostate Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Michael H. Antoni, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19990288; 1P50CA084944 (NIH)
Record Dates: First submitted 2022-08-02; First posted 2022-08-04 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Stress
Keywords: group therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive behavioral stress management group (Experimental): Participants received the cognitive behavioral stress management intervention for 10 weeks.
  Interventions: Behavioral: Cognitive behavioral stress management
- Health promotion group (Active Comparator): Participants received the health promotion group for one day.
  Interventions: Behavioral: Psychoeducational Control

INTERVENTIONS:
Behavioral: Cognitive behavioral stress management — Participants will receive in-person weekly stress management group sessions (3-8 participants) for two hours per week for ten weeks total. Each session will consist of a half hour of relaxation training and one and a half hours of stress management skill training, including coping effectiveness training, anger management, assertiveness training, and stress awareness.
  Arms: Cognitive behavioral stress management group
Behavioral: Psychoeducational Control — Participants will receive one four-hour seminar in-person groups (3-8 participants) of educational information related to prostate cancer and abbreviated psychological information provided in cognitive behavioral stress management.
  Arms: Health promotion group

SUMMARY:
The purpose of this study is to test a stress management program for men with early-stage prostate cancer.

ELIGIBILITY:
Inclusion criteria:

* Men who had undergone either a radical prostatectomy or radiation therapy (i.e., external beam or seed implant) for stage I or II prostate cancer in the preceding 18-months
* 50 years of age or older
* Ability to speak, read, and write in English
* Having a ninth grade reading level or greater
* Being free of cognitive impairment that would interfere with the study
* No active psychiatric symptoms in the previous three months.

Exclusion criteria:

* Previous history of non-skin cancer
* Have received adjuvant treatment, including hormone treatment, for prostate cancer

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 1999-06-22 (Actual); Primary Completion 2006-08-03 (Actual); Study Completion 2006-08-03 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Stress Management Abilities as measured by the Measure of Current Status Questionnaire | Baseline, up to 18 months
  The Measure of Current Status questionnaire is a 23-item questionnaire each scored on a range of 0-4. The total score ranges from 0-92 with the higher score corresponding to greater perceived abilities.
Change in post-traumatic event perceptions as measured by the Benefit Finding Scale questionnaire | Baseline, up to 18 months
  The Benefit Finding Scale questionnaire is a 17-item measure capturing perception of a traumatic event (e.g., cancer diagnosis for participants) with each item scored on a scale of 1 to 5. The total score ranges from 17-85 with the higher score corresponding to greater perceived benefit.
Change in optimism as measured by the Life Orientation Test - Revised questionnaire | Baseline, up to 18 months
  The Life Orientation Test - Revised questionnaire measures participant's optimism. The total score ranges from 0-24 with the higher score corresponding to greater levels of optimism.
Change in immune cell count | Baseline, up to 18 months
  Immune cell count (including T-cell (Cluster of Differentiation (CD) 3+) and T-helper cells (CD 3+ CD 4+) will be evaluated from blood samples. Both values will be evaluated in count per cubic millimeter.
Change in immune cell percentage | Baseline, up to 18 months
  Immune cell percentage (including T-cell (Cluster of Differentiation (CD) 3+) and T-helper cells (CD 3+ CD 4+) will be evaluated from blood samples. Both values evaluated in count per cubic millimeter over total cell count per cubic millimeter.
Change in natural killer cell percentage | Baseline, up to 18 months
  Natural killer cell (CD56+CD3-) percentage is evaluated from blood samples. Values are evaluated in count per cubic millimeter over total cell count per cubic millimeter.
Change in natural killer cell count | Baseline, up to 18 months
  Natural killer cell (CD56+CD3-) count is evaluated from blood samples. Values are evaluated in count per cubic millimeter.
Change in natural killer cell cytotoxicity as captured by activity percentage | Baseline, up to 18 months
  Natural killer cell (CD56+CD3-) cytotoxicity is evaluated from blood samples. Cells are stimulated through exposure to a reactive cell line and the percentage of cells active are counted and divided by total cells present per cubic millimeter.
Change in ratio of natural killer cell cytotoxicity as captured by Lytic Index | Baseline, up to 18 months
  Natural killer cell (CD56+CD3-) cytotoxicity is evaluated from blood samples. Cells are stimulated through exposure to a reactive cell line and quantified as the ratio of responsive to unresponsive cells required to kill 10% of the target cell line.
Change in count of natural killer cell cytotoxicity as captured by Kinetic Lytic Index | Baseline, up to 18 months
  Natural killer cell (CD56+CD3-) cytotoxicity is evaluated from blood samples. Cells are stimulated through exposure to a reactive cell line and incubated for four hours total. Kinetic lytic index is quantified as the count of targeted cells killed during incubation. An average count of these cells will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Antoni, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Penedo FJ, Molton I, Dahn JR, Shen BJ, Kinsinger D, Traeger L, Siegel S, Schneiderman N, Antoni M. A randomized clinical trial of group-based cognitive-behavioral stress management in localized prostate cancer: development of stress management skills improves quality of life and benefit finding. Ann Behav Med. 2006 Jun;31(3):261-70. doi: 10.1207/s15324796abm3103_8. PMID 16700640
- [Result] Traeger L, Penedo FJ, Benedict C, Dahn JR, Lechner SC, Schneiderman N, Antoni MH. Identifying how and for whom cognitive-behavioral stress management improves emotional well-being among recent prostate cancer survivors. Psychooncology. 2013 Feb;22(2):250-9. doi: 10.1002/pon.2074. Epub 2011 Sep 19. PMID 21932396
- [Result] Molton IR, Siegel SD, Penedo FJ, Dahn JR, Kinsinger D, Traeger LN, Carver CS, Shen BJ, Kumar M, Schneiderman N, Antoni MH. Promoting recovery of sexual functioning after radical prostatectomy with group-based stress management: the role of interpersonal sensitivity. J Psychosom Res. 2008 May;64(5):527-36. doi: 10.1016/j.jpsychores.2008.01.004. PMID 18440406
- [Derived] Walsh EA, Antoni MH, Popok PJ, Moreno PI, Penedo FJ. Effects of a randomized-controlled trial of cognitive behavioral stress management: Psychosocial adaptation and immune status in men with early-stage prostate cancer. Gen Hosp Psychiatry. 2022 Nov-Dec;79:128-134. doi: 10.1016/j.genhosppsych.2022.10.012. Epub 2022 Oct 27. PMID 36375341